CLINICAL TRIAL: NCT06922526
Title: Predictors of Tricuspid Regurgitation Progression and Adverse Outcomes in Different Pacing Modes
Brief Title: Pacemaker-related Tricuspid Regurgitation Progression and Long-term Outcomes
Status: Recruiting | Type: Observational
Sponsor: Haiyan Wang (Other)
Responsible Party: Sponsor-Investigator, Haiyan Wang, Director, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: SDYWZGKCJH2024030
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Tricuspid Regurgitation; Pacemaker
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Right ventricular pacing group
  Interventions: Device: Pacemaker implantation
- conduction system pacing group
  Interventions: Device: Pacemaker implantation
- biventricular pacing group
  Interventions: Device: Pacemaker implantation
- TR progression group
- non-TR progression group

INTERVENTIONS:
Device: Pacemaker implantation — Pacemaker implantation methods include right ventricular pacing, biventricular pacing, conduction system pacing
  Groups: Right ventricular pacing group; biventricular pacing group; conduction system pacing group

SUMMARY:
Tricuspid regurgitation (TR) is a common complication following cardiac implantable electronic device (CIED) implantation, with severe TR being associated with increased rates of heart failure hospitalization and all-cause mortality, significantly impairing patients' quality of life. With technological advancements, physiological pacing modalities have demonstrated superior clinical efficacy and safety profiles compared to conventional pacing methods.

This study aims to evaluate predictors of adverse outcomes and TR progression in CIED recipients under different pacing modalities, thereby providing clinical guidance for high-risk patients.

DETAILED DESCRIPTION:
This retrospective study analyzed patients undergoing pacemaker implantation from January 2015 to March 2025, stratified by pacing modality (right ventricular/conduction system/biventricular pacing) and TR progression (worsened [≥1-grade increase] vs non-worsened TR).

The protocol included: (1) 3D echocardiographic assessment of TR mechanisms, (2) quantitative fluoroscopic analysis of lead parameters (tension, mobility, angulation), (3) multivariable regression evaluating pacing modes and TR progression on clinical outcomes, and (4) documentation of device-related complications (lead dislodgement/infection) and heart failure rehospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. Patients with an implantable electronic heart device (CIEDs)
3. The patient underwent pacemaker implantation at Qianfoshan Hospital between 2015 and 2025

Exclusion Criteria:

1. Patients with severe tricuspid regurgitation or those who have undergone tricuspid valve surgery or interventional treatment prior to pacemaker implantation
2. Patients with severe valvular heart disease, congenital heart disease, or arrhythmias
3. Patients with single-chamber pacemakers or poor images

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after cardiac pacemaker implantation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Tricuspid regurgitation progression（Progression of tricuspid regurgitation ≥ grade 0.5） | Mean follow-up of 1 year
  Grading of tricuspid regurgitation severity:Grade 0: None
  Grade 0.5: Trace
  Grade 1: Mild
  Grade 1.5: Mild to moderate
  Grade 2: Moderate
  Grade 2.5: Moderate to severe
  Grade 3: Severe

SECONDARY OUTCOMES:
Heart Failure Readmission Rate After CIED Implantation | Mean follow-up of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Wang, MD, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoke U, Auger D, Thijssen J, Wolterbeek R, van der Velde ET, Holman ER, Schalij MJ, Bax JJ, Delgado V, Marsan NA. Significant lead-induced tricuspid regurgitation is associated with poor prognosis at long-term follow-up. Heart. 2014 Jun;100(12):960-8. doi: 10.1136/heartjnl-2013-304673. Epub 2014 Jan 21. PMID 24449717
- [Background] Li X, Fan X, Wang Q, Wang Z, Zhu H, Li H, Wang H, Liu Z, Yao Y. Tricuspid regurgitation following pacemaker implantation for bradycardia: a two-year study comparing different pacing strategies. Chin Med J (Engl). 2023 Oct 20;136(20):2508-2510. doi: 10.1097/CM9.0000000000002825. Epub 2023 Aug 31. No abstract available. PMID 37649400
- [Background] Li X, Zhu H, Fan X, Wang Q, Wang Z, Li H, Tao J, Wang H, Liu Z, Yao Y. Tricuspid regurgitation outcomes in left bundle branch area pacing and comparison with right ventricular septal pacing. Heart Rhythm. 2022 Jul;19(7):1202-1203. doi: 10.1016/j.hrthm.2022.03.005. Epub 2022 Mar 10. No abstract available. PMID 35278699